CLINICAL TRIAL: NCT03517241
Title: A Multimodal Approach Towards an Objective Assessment of Macular Function at Retinal and Cortical Levels
Brief Title: Objective Assessment of Macular Function at Retinal and Cortical Levels
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Markus Ritter, MD, Associate Professor, Medical University of Vienna
Other Study IDs: EK1816/2014
Record Dates: First submitted 2018-04-17; First posted 2018-05-07 (Actual); Last update posted 2018-05-07 (Actual); Status verified 2018-05

CONDITIONS: Macula; Degeneration, Congenital or Hereditary; Retina Disorder
MeSH Terms: conditions — Retinal Diseases | interventions — Magnetic Resonance Imaging; Tomography, Optical Coherence; Vision Tests

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Geographic atrophy secondary to AMD: 20 patients clinically diagnosed with geographic atrophy (GA) secondary to AMD.
  Interventions: Diagnostic Test: functional magnetic resonance imaging (fMRI); Diagnostic Test: Microperimetry (MP); Diagnostic Test: Optical coherence tomography (OCT); Diagnostic Test: Blue light fundus autofluorescence imaging (FAF); Diagnostic Test: Visual testing
- Stargards disease: 20 patients clinically and genetically diagnosed with Stargards disease (STGD)
  Interventions: Diagnostic Test: functional magnetic resonance imaging (fMRI); Diagnostic Test: Microperimetry (MP); Diagnostic Test: Optical coherence tomography (OCT); Diagnostic Test: Blue light fundus autofluorescence imaging (FAF); Diagnostic Test: Visual testing
- Branch retinal artery occlusion: 20 patients clinically diagnosed with branch retinal artery occlusion (BRAO)
  Interventions: Diagnostic Test: functional magnetic resonance imaging (fMRI); Diagnostic Test: Microperimetry (MP); Diagnostic Test: Optical coherence tomography (OCT); Diagnostic Test: Blue light fundus autofluorescence imaging (FAF); Diagnostic Test: Visual testing
- Full thickness macular hole: 20 patients clinically diagnosed with acute full thickness macular hole (FTMH) before and after macular surgery
  Interventions: Diagnostic Test: functional magnetic resonance imaging (fMRI); Diagnostic Test: Microperimetry (MP); Diagnostic Test: Optical coherence tomography (OCT); Diagnostic Test: Blue light fundus autofluorescence imaging (FAF); Diagnostic Test: Visual testing
- Healthy controls: 20 healthy control subjects. Visual acuity of 20/16- 20/32
  Interventions: Diagnostic Test: functional magnetic resonance imaging (fMRI); Diagnostic Test: Microperimetry (MP); Diagnostic Test: Optical coherence tomography (OCT); Diagnostic Test: Blue light fundus autofluorescence imaging (FAF); Diagnostic Test: Visual testing

INTERVENTIONS:
Diagnostic Test: functional magnetic resonance imaging (fMRI) — Retinotopic mapping using functional magnetic resonance imaging (fMRI) is based on MR images acquired with blood-oxygenation-level-dependent (BOLD) contrast to reveal areas of neuronal activity in the visual cortex
Diagnostic Test: Microperimetry (MP) — MP allows localized testing of retinal sensitivity of foveal, parafoveal and even more peripheral macular regions
Diagnostic Test: Optical coherence tomography (OCT) — Optical Coherence Tomography (OCT) is a non-invasive diagnostic technique that renders an in vivo cross sectional view of the retina.
Diagnostic Test: Blue light fundus autofluorescence imaging (FAF) — Fundus autofluorescence imaging (FAF), is a non-invasive diagnostic technique focusing on the fluorescent properties of pigments in the retina to generate images.
Diagnostic Test: Visual testing — Best-corrected visual acuity will be measured using Early Treatment Diabetic Retinopathy Study (ETDRS) charts. Reading acuity and reading speed will be examined using Radner Reading Charts. Reading acuity is measured in logRAD unit (= reading equivalent of logMAR) and in critical font size (critical reading size), reading speed is measured in words per minute (wpm). Contrast sensitivity will be determined using Pelli-Robson contrast sensitivity charts.

SUMMARY:
Research questions/hypotheses: About 15% of the population over 40 years of age are affected by diseases of the retina. Accurate measurement of the extent of visual field impairment is of highest importance for disease subtype diagnosis and severity classification. The current gold-standard approach for the assessment of macular sensitivity is microperimetry (MP) where the patient is asked to report whether or not visual stimuli presented at different positions within the visual field are detected. While this technique is a very straightforward approach and simple in its application, it is important to note that MP is psychophysical in nature and requires constantly high attentional performance of the patient throughout the examination period. As many patients suffering from retinal diseases are well over 65 years of age, they are unable to maintain such high levels of attention over longer periods and, thus, MP results may be biased. Retinotopic assessment using population receptive field (pRF) mapping based on functional magnetic resonance imaging (fMRI) offers an alternative by allowing for objective visual field testing, independent of patient performance. We have shown previously in healthy subjects that pRF allows for accurate detection of simulated central scotomata down to 2.35 degrees radius. Also, pilot data in patients with retinal scotomata showed strong correspondence between pRF and MP results, i.e. macular regions with reduced macular sensitivity and atrophy of outer retinal layers correlated well with pRF coverage maps showing reduced density of activated voxels. The aim of this project is to determine whether pRF mapping could serve as an alternative visual field testing method by: (1) assessing test-retest reproducibility of pRF and MP in clinical populations with stable retinal diseases (Stargardt disease, geographic atrophy) over a four-week period; (2) assessing visual field changes over a one-year period in patients suffering from acute retinal scotomata (branch retinal artery occlusions, full-thickness macular holes). All pRF mapping will be accompanied by MP measurements to allow for a direct comparison of the two techniques.

Scientific/scholarly innovation/originality of the project: The present project applies a novel approach for linking retinal function assessed with MP and pRF mapping in a representative patient population with acute and chronic retinal diseases. The project seeks to contribute to best practice methods for using fMRI to assess macular dysfunction both for documentation of the natural course of the disease and during therapy in a study setting.

Methods: fMRI uses pRF mapping to provide retinotopic data (pRF coverage maps) that are then correlated with the results of conventional ophthalmic testing including MP, visual acuity and contrast sensitivity testing, reading performance, optical coherence tomography and autofluorescence imaging.

ELIGIBILITY:
Inclusion Criteria:

* 20 patients clinically diagnosed with GA secondary to AMD.
* 20 patients clinically and genetically diagnosed with STGD.
* 20 patients clinically diagnosed with BRAO.
* 20 patients clinically diagnosed with acute FTMH before and after macular surgery.
* 20 healthy control subjects. Visual acuity of 20/16- 20/32

Exclusion Criteria:

* Presence of any other ophthalmological or neurological disease affecting visual function
* Cataract > grade 2 (according to lens opacities system)
* All routine exclusion criteria that apply to MRI scans including pacemakers, metallic implants, prostheses or coils, claustrophobia
* Pregnancy
* Dyslexia

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Consecutive enrollment from the Macular Disease Unit of the Dept. of Ophthalmology, Medical University of Vienna.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-05-15 (Estimated); Primary Completion 2020-03-16 (Estimated); Study Completion 2020-06-15 (Estimated)

PRIMARY OUTCOMES:
Correspondence between coverage maps originating from microperimetry and population-receptive field mapping of the primary visual cortex measured by functional magnetic resonance imaging. | 2 years
  Qualitative and quantitative assessment of the correspondence between conventional functional assessment of retinal scotomata (microperimetry) and population-receptive field (pRF) mapping of the primary visual cortex measured by functional magnetic resonance imaging in patients clinically diagnosed with geographic atrophy secondary to age-related macular degeneration, Stargardts disease, branch retinal artery occlusions and full thickness macular holes before and after macular surgery. The microperimetry test grid (retinal sensitivity measured in Decibel, dB) willl be correlated with the pRF coverage maps calculated from fMRI data. Each dot represents the centre of a receptive field of a single voxel and every pRF centre is associated with a 2D Gaussian which together constitute the coverage map. Correspondence between coverage maps will be quantified by calculating the matching coefficient.

SECONDARY OUTCOMES:
Correspondence between coverage maps originating from structural imaging (optical coherence tomography and autofluorescence imaging) and population-receptive field mapping of the primary visual cortex measured by functional magnetic resonance imaging. | 2 years
  Qualitative and quantitative assessment of the correspondence between conventional structural assessment of retinal scotomata (optical coherence tomography and autofluorescence imaging) and population-receptive field (pRF) mapping of the primary visual cortex measured by functional magnetic resonance imaging in patients clinically diagnosed with geographic atrophy secondary to age-related macular degeneration, Stargardts disease, branch retinal artery occlusions and full thickness macular holes before and after macular surgery. The retinal layer thickness maps (measured in micometer, µm) willl be correlated with the pRF coverage maps calculated from fMRI data. Each dot represents the centre of a receptive field of a single voxel and every pRF centre is associated with a 2D Gaussian which together constitute the coverage map.Correspondence between coverage maps will be quantified by calculating the matching coefficient.
Reproducibility assessment | 1 year
  Reproducibility of population-receptive field mapping of the primary visual cortex and of conventional ophthalmic assessment (microperimetry, visual acuity and contrast sensitivity testing, reading performance, optical coherence tomography and autofluorescence imaging) in patients with retinal scotomata secondary to Stargardt disease and geographic atrophy compared with normal control participants with artificial scotomata.

IPD SHARING:
Plan to Share IPD: No